CLINICAL TRIAL: NCT00456118
Title: Study of the Role of Tissular Maternofetal Alloimmunization in Placentation Pathologies
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I06014
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2009-05

CONDITIONS: Recurrent Pregnancy Losses; Preeclampsia; Intervillositis
Keywords: recurrent pregnancy losses; preeclampsia; intervillositis; maternofetal alloimmunization
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- repeated miscarriages: 60 womens for repeated miscarriages will be included
- Preeclampsia: 70 women for pre-eclampsia will be included
- intervillites: 20 women for intervillites will be included

SUMMARY:
Justification:

We have recently demonstrated that maternofetal alloimmunization was not limited to blood cells: maternal alloimmunization against a glomerular podocyte antigen expressed by the placenta can induce neonatal membranous glomerulonephritis.

Early recurrent pregnancy losses, preeclampsia and intervillositis are obstetrical pathologies which share an anomaly of placentation. Pathophysiology of these diseases is not yet fully understood; nevertheless the hypothesis of an incompatibility between mother and child is often mentioned. The aim of this project is to detect and study the cases of recurrent pregnancy losses, preeclamspia and intervillositis which could be induced by tissular maternofetal alloimmunization.

Materials and methods:

Patients suffering from recurrent pregnancy losses of unknown origin, preeclamspia or intervillositis will be included in this project. Mothers' sera will be studied by indirect immunofluorescence and Western Blot on placental biopsies from different origins and gestational ages. This stage will enable us to detect possible maternal allo-antibodies. After detecting and revealing antibodies, nature of the target antigen will be identified by immunoprecipitation of placental extracts, using the positive sera. Immunoprecipitation will be followed by a mass spectrometry analysis of detected proteins.

Expected results:

This study will enable us:

* to detect new cases of tissular maternofetal alloimmunization
* to improve our knowledge of mechanisms leading to anomalies of placentation
* to carry out a specific, preventive therapeutic approach for cases induced by tissular alloimmunization.

Key words:

Recurrent pregnancy losses, Preeclampsia, Intervillositis, maternofetal alloimmunization.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent pregnancy losses : patient having or having suffered from at least 3 consecutive, unexplained recurrent pregnancy losses, during the first 3 months of pregnancy, with the same paerson/man.
* Preeclampsia : blood pressure > 140/90 mm Hg ; proteinuria > 0,3 g/ 24 h
* Intervillositis : patient suffering or having suffered from intervillositis

Exclusion Criteria:

* Recurrent pregnancy losses : uterine pathology, endocrine pathology, autoimmune pathology, coagulation and hemostasis pathology, karyotype anomaly.
* Preeclampsia : pre-existing high blood pressure, pre-existing diabetes, pre-existing renal disease, antiphospholipid antibodies syndrome
* Intervillositis : intervillositis with villositis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Neonatal pathologies can be caused by an alloimmunisation maternal fetal tissue, it's conceivable that certain pathologies. Obstetrics may be part of the same mechanism. Among these pathologies placentaires, for whom a "maternal-fetal incompatibility" is often mentioned, could be secondary to tissue alloimmunization against antigens independent of the immune system
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GUIGONIS, MD, Principal Investigator — University Hospital, Limoges
Locations (7):
- France (7):
  - Bordeaux University Hospital, Bordeaux
  - LIMOGES University Hospital, Limoges
  - Saint Antoine Hospital, Paris
  - Tenon Hospital, Paris
  - Trousseau Hospital, Paris
  - South Reunion Hospital, Saint-Pierre
  - Toulouse University Hospital, Toulouse